CLINICAL TRIAL: NCT05145725
Title: Instrumented POsterolateral Arthrodesis for Adolescent Idiopathic Scoliosis: Observational Study
Brief Title: Instrumented POsterolateral Arthrodesis for Adolescent Idiopathic Scoliosis
Acronym: APOSIA
Status: Recruiting | Type: Observational
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other); Asociación European Spine Study Group (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-A03069-30
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Scoliosis; Adolescence; Arthrodesis
MeSH Terms: conditions — Scoliosis; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic scoliosis in adolescents requiring surgery
  Interventions: Behavioral: Quality of life questionnaires

INTERVENTIONS:
Behavioral: Quality of life questionnaires — Different questionnaires to fill : SRS-22r, SF-36 score, TAPS, KIDSCREEN10

SUMMARY:
The study population concerns adolescent patients with idiopathic scoliosis which requires surgical management and who have a longer waiting period of 6 months.

The aim of this study is to research the predictive factors of an improvement in the quality of life of adolescents who have had surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 12 and 20 years old
* Scoliosis in adolescents for whom surgery has been proposed based on radiological criteria (Cobb angle> 25 ° for thoracolumbar and lumbar scoliosis,> 35 ° for thoracic scoliosis and> 40 ° for double major scoliosis)
* Patient affiliated or beneficiary of a social security scheme or attached to a beneficiary of a social security scheme
* Patient and legal representative having been informed and not opposing this research

Exclusion Criteria:

* Patient over 20 years old
* Non-surgical scoliosis
* Refusal to participate in the study by the child or parents

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents between 12 and 20 years old, suffering from scoliosis. Surgery has been proposed to them. 150 patients are French over the 866 patients.
Sampling Method: Probability Sample
Enrollment: 866 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2028-03-18 (Estimated); Study Completion 2036-03-18 (Estimated)

PRIMARY OUTCOMES:
Factors associated with an improvement in the SRS-22r score | 1 year
  Factors associated with an improvement in the SRS-22r score, 1 year after surgery, will be sought among the initial characteristics (before surgery) and within 3 months after surgery. An improvement in SRS-22r score is defined as an increase in the total score at 1 year of at least 10% from value.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du dos, Bruges, France